CLINICAL TRIAL: NCT04431154
Title: Financial Incentives to Promote Linkage to Care and Viral Suppression Following HIV Testing: a Randomized Controlled Trial
Brief Title: Incentives to Promote Sustained Linkage to HIV Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Wits Reproductive Health and HIV Institute (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: HSTAR013
Record Dates: First submitted 2020-06-10; First posted 2020-06-16 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Human Immunodeficiency Virus; HIV/AIDS
Keywords: HIV self-testing; Behavioral sciences; Financial incentives; Viral suppression
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Individuals who report results of a positive HIV test will be randomized 1:1 to the intervention (incentives) or control (no incentives) arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Usual care (No Intervention): Participants randomized to this arm will receive the standard of care (SOC) following the STAR program protocol in various sites in Johannesburg. This will include provision of an HIV self-screening test kit, the standard linkage officer follow-up call following report of a positive HIVSS test and an invitation to i) participate in study visit 1 to have their positive HIVSS result confirmed and complete blood collection for viral load PCR testing and to ii) participate in study visit 2 at 6 months for Viral Load PCR. Individuals with a positive HIV test result from another Ezintsha study or an affiliated clinic will also be invited to participate in study visit 1 for baseline viral load PCR testing.
- Experimental: Incentives and linkage promotion (Experimental): Participants randomized to this arm will receive the same standard HIV self-screen test kit and linkage officer follow-up call including the invitation to i) participate in study visit 1 and ii) study visit 2. In addition, they will receive a financial incentive if they complete a confirmatory HIV test at visit 1 and if they demonstrate viral suppression at study visit 2, approximately 6 months after positive HIVSS result. They will also receive monthly reminders and incentives to pick up HIV medication. Individuals with a positive HIV test result from another Ezintsha study or an affiliated clinic will also be invited to participate in study visit 1 for baseline viral load PCR testing.
  Interventions: Behavioral: Provision of HIV self-screen kit with incentives and linkage promotion

INTERVENTIONS:
Behavioral: Provision of HIV self-screen kit with incentives and linkage promotion — This arm will receive a HIV self-screen kit and additional incentives to promote adherence and linkage to care
  Arms: Experimental: Incentives and linkage promotion

SUMMARY:
This study aims to test if small incentives promote linkage to care and 6-month viral suppression among individuals recently tested for HIV at selected sites within Johannesburg, South Africa. Individuals who obtain a reactive HIV test result will be randomized to receive either the standard of care (SOC) for linkage to care or to receive financial incentives for confirmatory testing, linkage to care and viral suppression.

DETAILED DESCRIPTION:
This study is in collaboration with Ezintsha, a sub-division of Wits Reproductive Health and HIV Institute (WRHI) in South Africa. This study will leverage on the existing research infrastructure of Ezintsha, including, HIVSS testing through the STAR initiative (Self-Test Africa), as well as HIV positive persons identified through other Ezintsha research studies and at Eztinsha affiliated health clinics.

This study will use a randomized trial design to test the effectiveness of incentives to increase confirmatory testing, linkage to care and viral suppression. The aim of this study is to determine whether HIV-infected men and women are more likely to achieve or maintain HIV virologic suppression if offered financial incentives vs. no incentives (standard of care).

Individuals who report receiving a reactive HIVSS test result on the STAR programme, or a HIV reactive test in another research study or at a affiliated clinic, will be randomized into one of two groups: a) a control group that receives the standard of care (SOC) for linkage to care; and b) an intervention group that receives financial incentives for confirmatory testing, linkage to care, and viral suppression.

ELIGIBILITY:
Inclusion Criteria:

* Reported HIV positive
* Have a personal and/or valid phone number, that will remain active for 6 months
* Have a phone with WhatsApp, or text message feature
* Understand the Informed Consent form

Exclusion Criteria:

* Unwilling to provide informed consent
* Any condition which would make the participant unsuitable or unsafe for enrollment, i.e. being unable to see or read by forgetting to bring reading glasses, being intoxicated or acute sickness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Viral suppression at 6 months | approximately 6 months
  Viral suppression (plasma HIV RNA <400 copies/mL) at approximately 6 months after a positive HIV result

SECONDARY OUTCOMES:
Confirmatory testing | approximately 4 weeks
  Laboratory HIV confirmatory testing within approximately 4 weeks for participants with a positive HIV self-screening result.
ART initiation | approximately 4 weeks
  ART initiation within approximately 4 weeks after for those newly diagnosed with HIV

CONTACTS AND LOCATIONS:
Overall Officials: Harsha Thirumurthy, PhD, Principal Investigator — University of Pennsylvania; Mohammed Majam, MBA, Principal Investigator — Ezintsha, sub-division of Wits Reproductive Health and HIV Institute
Locations (1):
- Ezintsha Clinical Research Center, Johannesburg, Gauteng, South Africa